CLINICAL TRIAL: NCT03258437
Title: A 12-week, Multi-center, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Allium Cepa L. and Cuscuta Chinensis Lam. Extract Mixtures (DA-9401) on Improvement of Sperm Motility
Brief Title: Efficacy and Safety of DA-9401 on Improvement of Sperm Motility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean Society for Sexual Medicine and Andrology (Other)
Responsible Party: Principal Investigator, Park Jong Kwan, Principal Investigator, Chonbuk National University Hospital, Urology, Korean Society for Sexual Medicine and Andrology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DA-9401-SM
Record Dates: First submitted 2017-07-05; First posted 2017-08-23 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Spermatocele
Keywords: sperm motility, Clinical Trial , DA-9401
MeSH Terms: conditions — Spermatocele | interventions — DA-9401

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA-9401 (Experimental): capsules (4cap/d, 2.16 g/d) for 12 weeks.
  Interventions: Dietary Supplement: DA-9401
- Placebo (Placebo Comparator): Placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DA-9401
  Other Names: capsules (4cap/d, 2.16 g/d) for 12 weeks.
  Arms: DA-9401
Dietary Supplement: Placebo — Placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Allium cepa L. and Cuscuta chinensis Lam. Extract Mixtures (DA-9401) on improvement of sperm motility.

DETAILED DESCRIPTION:
This study was a 12 weeks, multi-center, randomized, double-blind, placebo-controlled human trial. Twenty subjects were randomly divided into Allium cepa L. and Cuscuta chinensis Lam. Extract Mixtures (DA-9401) or a placebo group. sperm motility profiles before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-55 years
* sperm motility 40~69%

Exclusion Criteria:

* History of alcohol or substance abuse
* Participation in any other clinical trials within past 1 months
* intense constipation

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Changes of Sperm motility | 12 weeks
  Changes of sperm profile were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of Sperm count | 12 weeks
  Changes of Sperm count(X10^6(M)/ml) profile were assessed before and after the intervention
Changes of Ejaculated volume | 12 weeks
  Changes of Ejaculated volume(ml) profile were assessed before and after the intervention
Changes of Sperm morphology | 12 weeks
  Changes of Sperm morphology(%) profile were assessed before and after the intervention
Changes of Ejaculated pH | 12 weeks
  Changes of Ejaculated pH profile were assessed before and after the intervention
Changes of hormone(Total testosterone, FSH, LH) | 12 weeks
  Changes of hormone{Total testosterone(ng/ml), FSH and LH(mlU/ml)} profile were assessed before and after the intervention
Changes of IIEF(International Index of Erectile Function) | 12 weeks
  Changes of questionnaire profile were assessed before and after the intervention
Changes of MFS(Multidimensional Fatigue Scale) | 12 weeks
  Changes of questionnaire profile were assessed before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital of urology, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided